CLINICAL TRIAL: NCT02006758
Title: EnligHTN European Observational Study
Brief Title: Observational Study of the EnligHTN Renal Denervation System in Europe
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CV-12-064-EU-HT
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-08

CONDITIONS: Uncontrolled Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Uncontrolled hypertension patients: The study will enroll 500 patients planned to undergo a renal denervation procedure (with the 'EnligHTN™ Renal Denervation System') for the treatment of their uncontrolled hypertension.
  Interventions: Device: EnligHTN™ Renal Denervation System

INTERVENTIONS:
Device: EnligHTN™ Renal Denervation System — The EnligHTN™ Renal Denervation System is designed to deliver radiofrequency (RF) energy to the renal nerves to achieve targeted denervation. The system consists of the EnligHTN™ RF Ablation Generator (generator), the EnligHTN™ Renal Artery Ablation Catheter (ablation catheter), and the EnligHTN™ Guiding Catheter (optional).

SUMMARY:
The purpose of this observational study is to further evaluate the safety and performance of the EnligHTN™ Renal Denervation System in the treatment of participants with uncontrolled hypertension in clinical routine practice.

DETAILED DESCRIPTION:
The EnligHTN European Observational study is designed to collect more data, critical to the benefit of the therapy, within a clinical routine setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject is planned to undergo a renal denervation procedure for the treatment of hypertension
* Subject is ≥18 years of age at time of consent
* Subject must be able and willing to provide written informed consent
* Subject must be able and willing to comply with the required follow-up schedule
* Subject has office SBP ≥ 140 mmHg
* Subject has established hypertension (diagnosed ≥12 months prior to baseline) and is on a guideline based drug regimen at a stable (≥ 14 days) and a fully tolerated dose consisting of ≥3 anti-hypertensive medications (including 1 diuretic)

Exclusion Criteria:

* Subject has known significant renovascular abnormalities such as renal artery stenosis > 30%
* Subject has undergone prior renal angioplasty, renal denervation, indwelling renal stents, and/or abdominal aortic stent grafts
* Subject has a history of hemodynamically significant valvular heart disease
* Subject has blood clotting abnormalities
* Subject life expectancy is < 12 months, as determined by the Study Investigator
* Subject is participating in another clinical study which has the potential to impact his/her hypertension management (pharmaceutical/ device/ homeopathic)
* Subject is pregnant, nursing, or of childbearing potential and is not using adequate contraceptive methods
* Subject has active systemic infection
* Subject has known renal arteries with diameter(s) < 4 mm
* Subject has an estimated GFR <45 mL/min per 1.73 m2 using the Modification of Diet in Renal Disease (MDRD) formula
* Subject had a renal transplant or is awaiting a renal transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uncontrolled hypertension
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2013-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Diaz, MD, Principal Investigator — Hospital Juan Ramon Jimenez, Huelva, Spain
Locations (13):
- Hôpital Civil Marie Curie, Lodelinsart, Hainaut, Belgium
- North Estonia Medical Centre, Tallinn, Harjuma, Estonia
- Italy (4):
  - Dr. Gianluigi Patelli, Alzano Lombardo, Lombardy
  - Instituto Clinico Citta Studi, Milan, Lombardy
  - Policlinico San Marco, Osio Sotto, Lombardy
  - Clinica San Gaudenzio, Novara, Peimonte
- Hospital de Santa Cruz, Carnaxide, Lisbon District, Portugal
- Spain (5):
  - Hospital Juan Ramon Jimenez, Huelva, Andalusia
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hopspital Infanta Cristina, Badajoz
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Xeral-Cies de Vigo, Vigo
- Craigavon Area Hospital, Portadown, Nirelnd, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Uncontrolled Hypertension Participants: Renal denervation procedure with EnligHTN system for the treatment of uncontrolled hypertension
Period: Overall Study
Arm/Group | Uncontrolled Hypertension Participants
Started | 68 (Total number of enrolled participants)
Underwent Renal Denervation | 67 (Underwent renal denervation)
1-month Follow up | 66 (1-month follow up completed)
6-month Follow up | 60 (6-month follow up completed)
12-month Follow up | 55 (12-month follow up completed)
Completed | 55
Not Completed | 13
Not completed — Protocol Violation | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 4
Not completed — Procedurally excluded | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: 67 participants underwent renal denervation; 1 participant was excluded because of inclusion criteria violation
Groups:
- Uncontrolled Hypertension Participants: Renal denervation procedure with the EnligHTN System for the treatment of uncontrolled hypertension
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant was excluded due to inclusion criteria violation
  years
    number analyzed (Participants) | 67
    (all) | 59.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant was excluded due to inclusion criteria violation
  Participants
    number analyzed (Participants) | 67
    Female | 30
    Male | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 11
  Estonia | 3
  Italy | 27
  Portugal | 5
  Spain | 16
  United Kingdom | 6
Physical Assessment - Weight [Mean (Standard Deviation); unit: kg] — Population: 1 participant was excluded due to inclusion criteria violation
  kg
    number analyzed (Participants) | 67
    (all) | 88.8 (19.3)
Physical Assessment - Height [Mean (Standard Deviation); unit: cm] — Population: 1 subject was excluded due to inclusion criteria violation
  cm
    number analyzed (Participants) | 67
    (all) | 169.8 (10.0)
Physical assessment - Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: 1 participant was excluded due to inclusion criteria violation
  kg/m^2
    number analyzed (Participants) | 67
    (all) | 30.5 (5.0)
Hypertension (HTN) [Mean (Standard Deviation); unit: years] — Population: Data were not collected for all participants.
  years
    Years since HTN diagnosis: number analyzed (Participants) | 49
    Years since HTN diagnosis | 12.8 (11.5)
    Years since subject was on anti-HTN meds: number analyzed (Participants) | 35
    Years since subject was on anti-HTN meds | 11.1 (11.8)
Renal artery atherosclerosis [Count of Participants; unit: Participants] — Population: 1 participant was excluded due to inclusion criteria violation
  Participants
    number analyzed (Participants) | 67
    (all) | 2
Renal artery atherosclerosis percentage [Mean (Standard Deviation); unit: percentage (%)] — Population: 2 participants had renal artery atherosclerosis, of which both were located on the right side.
  percentage (%)
    Percentage (%) of atherosclerosis on the right: number analyzed (Participants) | 2
    Percentage (%) of atherosclerosis on the right | 25 (0.0)
    Percentage (%) of atherosclerosis on the left: number analyzed (Participants) | 2
    Percentage (%) of atherosclerosis on the left | NA (NA) — 2 participants had renal artery atherosclerosis, of which both were located on the right side.
Renovascular Hypertension [Count of Participants; unit: Participants] — Population: 1 participant was excluded due to inclusion criteria violation
  Participants
    number analyzed (Participants) | 67
    (all) | 0
Other Renal Disease [Count of Participants; unit: Participants] — Population: 1 participant was excluded due to inclusion criteria violation
  Participants
    number analyzed (Participants) | 67
    (all) | 11
Cardiovascular History [Count of Participants; unit: Participants] — Population: 1 participant was excluded because of inclusion criteria violation.
  Participants
    None: number analyzed (Participants) | 67
    None | 43
    Myocardial Infarction: number analyzed (Participants) | 67
    Myocardial Infarction | 4
    Coronary Artery Disease: number analyzed (Participants) | 67
    Coronary Artery Disease | 14
    Coronary Artery Bypass Graft: number analyzed (Participants) | 67
    Coronary Artery Bypass Graft | 2
    Percutaneous Coronary Intervention: number analyzed (Participants) | 67
    Percutaneous Coronary Intervention | 10
    Abdominal Aortic Aneurysm: number analyzed (Participants) | 67
    Abdominal Aortic Aneurysm | 0
    Valvular Disease: number analyzed (Participants) | 67
    Valvular Disease | 3
    Arrhythmias: number analyzed (Participants) | 67
    Arrhythmias | 6
    Cardiomyopathy: number analyzed (Participants) | 67
    Cardiomyopathy | 9
Neurological history [Count of Participants; unit: Participants] — Population: 1 participant was excluded due to inclusion criteria violation
  Participants
    number analyzed (Participants) | 67
    None | 60
    Cerebrovascular accident | 2
    Other | 5
Additional Medical History [Count of Participants; unit: Participants] — Population: 1 participant was excluded due to inclusion criteria violation
  Participants
    Hyperlipidemia: number analyzed (Participants) | 67
    Hyperlipidemia | 27
    Diabetes: number analyzed (Participants) | 67
    Diabetes | 25
    Smoker: number analyzed (Participants) | 67
    Smoker | 21
    Significant Alcohol intake: number analyzed (Participants) | 67
    Significant Alcohol intake | 5
Office Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data were not collected for all participants.
  mmHg
    Systolic Blood Pressure: number analyzed (Participants) | 66
    Systolic Blood Pressure | 163.7 (22.5)
    Diastolic Blood Pressure: number analyzed (Participants) | 66
    Diastolic Blood Pressure | 90.3 (15.2)
Ambulatory Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data were not collected for all participants
  mmHg
    24 Hour Systolic Blood Pressure: number analyzed (Participants) | 35
    24 Hour Systolic Blood Pressure | 155.0 (16.9)
    24 Hour Diastolic Blood Pressure: number analyzed (Participants) | 35
    24 Hour Diastolic Blood Pressure | 86.6 (14.7)
    Day time Systolic Blood Pressure: number analyzed (Participants) | 35
    Day time Systolic Blood Pressure | 158.1 (17.1)
    Day time Diastolic Blood Pressure: number analyzed (Participants) | 35
    Day time Diastolic Blood Pressure | 89.2 (14.9)
    Night time Systolic Blood Pressure: number analyzed (Participants) | 35
    Night time Systolic Blood Pressure | 149.6 (23.6)
    Night time Diastolic Blood Pressure: number analyzed (Participants) | 35
    Night time Diastolic Blood Pressure | 80.5 (16.1)
Heart Rate [Mean (Standard Deviation); unit: bpm (beats per minute)] — Population: Data were not collected for all participants
  bpm (beats per minute)
    Office Heart Rate: number analyzed (Participants) | 65
    Office Heart Rate | 69.4 (11.7)
    24-Hour Ambulatory Heart Rate: number analyzed (Participants) | 31
    24-Hour Ambulatory Heart Rate | 67.7 (12.1)
    Day time Ambulatory Heart Rate: number analyzed (Participants) | 30
    Day time Ambulatory Heart Rate | 70.3 (13.5)
    Night time Ambulatory Heart Rate: number analyzed (Participants) | 30
    Night time Ambulatory Heart Rate | 64.2 (13.6)
Participants on stable anti-HTN medication prior to enrollment [Count of Participants; unit: Participants] — Population: 1 participant was excluded due to inclusion criteria violation
  Participants
    number analyzed (Participants) | 67
    (all) | 67
Number of anti-HTN medications participant currently takes [Mean (Standard Deviation); unit: medications] — Population: 1 participant was excluded due to inclusion criteria violation
  medications
    number analyzed (Participants) | 67
    (all) | 4.3 (1.0)
Antiarrhythmic Medication currently being taken [Count of Participants; unit: Participants] — Please note: Same participant may be on multiple different medications, and counted in each category. Population: Antihypertensive medication usage information was available for all enrolled participants
  Participants
    ACE/angiotensin 2 receptor/direct renin inhibitors | 48
    Beta blockers | 42
    Calcium Channel Blocker | 48
    Diuretics | 61
    Other hypertensive medication | 40
Serum creatinine concentration [Mean (Standard Deviation); unit: umol/L] — Population: Data were not collected for all participants
  umol/L
    number analyzed (Participants) | 63
    (all) | 86.1 (27.9)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min per 1.73 m^2] — Population: Data were not collected for all participants
  mL/min per 1.73 m^2
    number analyzed (Participants) | 53
    (all) | 79.1 (24.5)
Urine Albumin to Creatinine Ratio [Mean (Standard Deviation); unit: mg/g] — Population: Data were not collected for all participants
  mg/g
    number analyzed (Participants) | 12
    (all) | 89.6 (235)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Office Systolic Blood Pressure at 6 Months
Time Frame: Baseline and 6 months
Population: 58 out of 67 participants analyzed for primary outcome measure of office systolic blood pressure at 6 months.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 58
mmHg | -13.6 (29.2)

2. Secondary Outcome: Assessment of Peri-procedural Adverse Events up Until 30 Days Post Procedure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 67
Participants
  Back Pain | 1
  Renal Artery Stenosis | 1
  Urinary Tract Infection | 1
  Viral Syndrome | 1

3. Secondary Outcome: Mean Change in Office Systolic Blood Pressure at 1 Month
Time Frame: Baseline and 1 month
Population: 61 out of 67 participants were analyzed for mean reduction in office Systolic Blood Pressure at 1 month.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 61
mmHg | -13.0 (28.2)

4. Secondary Outcome: Mean Change in Office Diastolic Blood Pressure at 1 Month
Time Frame: Baseline and 1 month
Population: 61 out of 67 analyzed for mean change in office Diastolic Blood Pressure at 1 month
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Uncontrolled Hypertension Patients: Renal denervation procedure with EnligHTN system for the treatment of uncontrolled hypertension
Arm/Group | Uncontrolled Hypertension Patients
Number analyzed (Participants) | 61
mmHg | -4.6 (16.7)

5. Secondary Outcome: Mean Change in Ambulatory Systolic Blood Pressure at 1 Month
Time Frame: Baseline and 1 month
Population: 23 out of 67 participants analyzed for mean change in ambulatory Systolic Blood Pressure at 1 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 23
mmHg | -6.8 (18.2)

6. Secondary Outcome: Mean Change in Ambulatory Diastolic Blood Pressure at 1 Month
Time Frame: Baseline and 1 month
Population: 23 out of 67 participants analyzed for mean change in ambulatory Diastolic Blood Pressure at 1 month.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 23
mmHg | -3.6 (9.7)

7. Secondary Outcome: Percentage of Subjects Achieving Office Systolic Blood Pressure < 140 mmHg at 1 Month
Time Frame: 1 month
Population: 62 out of 67 participants analyzed for percentage of subjects achieving office Systolic Blood Pressure < 140 mmHg at 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 62
Participants | 24

8. Secondary Outcome: Renal Function Change Based on eGFR (Estimated Glomerular Filtration Rate) at 6 Months
Time Frame: Baseline and 6 months
Population: 48 out of 67 analyzed for renal function change based on eGFR at 6 months.
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 48
mL/min per 1.73 m^2 | -1.0 (21.3)

9. Secondary Outcome: Renal Function Change Based on eGFR (Estimated Glomerular Filtration Rate) at 12 Months
Time Frame: Baseline and 12 months
Population: 38 out of 67 analyzed for renal function change based on eGFR at 12 months.
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 38
mL/min per 1.73 m^2 | -2.2 (21.1)

10. Secondary Outcome: Renovascular Safety at 6 Months (Renal Artery Stenosis)
Description: Assessment of renovascular safety as measured by new renal artery stenosis or aneurysm at the site of ablation.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 67
Participants | 1

11. Secondary Outcome: Mean Change in Office Systolic Blood Pressure at 12 Months
Time Frame: Baseline and 12 months
Population: 54 out of 67 participants analyzed for mean change in office Systolic Blood Pressure at 12 months.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 54
mmHg | -13.8 (24.7)

12. Secondary Outcome: Mean Change in Office Diastolic Blood Pressure at 6 Months
Time Frame: Baseline and 6 months
Population: 58 out of 67 participants analyzed for mean change in office Diastolic Blood Pressure at 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 58
mmHg | -6.7 (17.6)

13. Secondary Outcome: Mean Change in Office Diastolic Blood Pressure at 12 Months
Time Frame: Baseline and 12 months
Population: 54 out of 67 participants analyzed for mean change in office Diastolic Blood Pressure at 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 54
mmHg | -7.1 (16.1)

14. Secondary Outcome: Mean Change in Ambulatory Systolic Blood Pressure at 6 Months
Time Frame: Baseline and 6 months
Population: 29 out of 67 participants analyzed for mean change in ambulatory Systolic Blood Pressure at 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 29
mmHg | -10.8 (13.7)

15. Secondary Outcome: Mean Change in Ambulatory Systolic Blood Pressure at 12 Months
Time Frame: Baseline and 12 months
Population: 25 out of 67 participants analyzed for mean change in ambulatory Systolic Blood Pressure at 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 25
mmHg | -6.4 (19.5)

16. Secondary Outcome: Mean Change in Ambulatory Diastolic Blood Pressure at 6 Months
Time Frame: Baseline and 6 months
Population: 29 out of 67 participants analyzed for mean change in ambulatory Diastolic Blood Pressure at 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 29
mmHg | -5.6 (7.1)

17. Secondary Outcome: Mean Change in Ambulatory Diastolic Blood Pressure at 12 Months
Time Frame: Baseline and 12 months
Population: 25 out of 67 participants analyzed for mean change in ambulatory Diastolic Blood Pressure at 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 25
mmHg | -4.2 (10.4)

18. Secondary Outcome: Percentage of Participants Achieving Office Systolic Blood Pressure < 140 mmHg at 6 Months
Time Frame: 6 months
Population: 59 out of 67 participants were analyzed for percentage of subjects achieving office Systolic Blood Pressure < 140 mmHg at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 59
Participants | 21

19. Secondary Outcome: Percentage of Participants Achieving Office Systolic Blood Pressure < 140 mmHg at 12 Months
Time Frame: 12 months
Population: 55 out of 67 participants were analyzed for percentage of subjects achieving office Systolic Blood Pressure < 140 mmHg at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 55
Participants | 19

20. Post Hoc Outcome: Serum Creatinine Concentration at 6 Months
Time Frame: 6 months
Population: 55 out of 67 analyzed for serum creatinine concentration at 6 months.
Measure: Mean (Standard Deviation); unit: umol
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 55
umol | 227.9 (1013.1)

21. Post Hoc Outcome: Serum Creatinine Concentration at 12 Months
Time Frame: 12 months
Population: 46 out of 67 analyzed for serum creatinine concentration at 6 months.
Measure: Mean (Standard Deviation); unit: umol
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 46
umol | 90.2 (29.5)

22. Post Hoc Outcome: Urine Albumin to Creatinine Ratio at 6 Months
Time Frame: 6 months
Population: 17 out of 67 analyzed for serum creatinine concentration at 6 months.
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 17
mg/g | 212.8 (635.1)

23. Post Hoc Outcome: Urine Albumin to Creatinine Ratio at 12 Months
Time Frame: 12 months
Population: 14 out of 67 analyzed for serum creatinine concentration at 6 months.
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 14
mg/g | 179.0 (373.1)

24. Post Hoc Outcome: Number of Anti-hypertensive Medications Participant Currently Takes at 12 Months
Time Frame: 12 months
Population: 55 out of 67 participants were analyzed for number of anti-hypertensive medications taken at 12 months
Measure: Mean (Standard Deviation); unit: number of medications
Arm/Group | Uncontrolled Hypertension Participants
Number analyzed (Participants) | 55
number of medications | 3.7 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 12 months.
Arm/Group | Uncontrolled Hypertension Participants
All-Cause Mortality (participants affected / at risk) | 1/68
Serious Adverse Events (participants affected / at risk) | 8/68
Other Adverse Events (participants affected / at risk) | 5/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uncontrolled Hypertension Participants (N=68)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Myocardial Ischemia (Cardiac disorders) | 1 (1)
Renal Artery Stenosis (Vascular disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sustained Atrial Fibrillation (Cardiac disorders) | 1 (1)
Viral Syndrome (Infections and infestations) | 1 (1)
VASC Vessel Stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uncontrolled Hypertension Participants (N=68)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Arterial Hypertension/Hypertension (Cardiac disorders) | 1 (1)
Bacterial Infections of the Skin (Infections and infestations) | 1 (1)
Drug Side Effect (General disorders) | 1 (1)
Urinary Tract Infections (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT02006758/Prot_SAP_000.pdf